CLINICAL TRIAL: NCT02227667
Title: Phase II Study to Evaluate the Efficacy of MEDI4736 in Immunological Subsets of Advanced Colorectal Cancer
Brief Title: Evaluate the Efficacy of MEDI4736 in Immunological Subsets of Advanced Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: MedImmune LLC (Industry); AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14-109
Record Dates: First submitted 2014-07-17; First posted 2014-08-28 (Estimated); Results first posted 2021-06-18 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2021-05

CONDITIONS: Advanced Colorectal Cancer
Keywords: MEDI4736; 14-109
MeSH Terms: interventions — durvalumab

ARMS (1):
- Patients with Advanced Colorectal Cancer (Experimental): This will be a Simon two-stage design, single arm, phase II study. All subjects will receive MEDI4736 via IV infusion. Subjects will continue treatment for 12 months, or until progression of disease, initiation of alternative cancer therapy, unacceptable toxicity, or other reasons to discontinue treatment occur. Following the 12-month treatment period, subjects without evidence for progressive disease or other reason to discontinue treatment will be monitored without further treatment. Upon evidence of PD (with or without confirmation according to RECIST 1.1) during the monitoring period, administration of MEDI4736 may resume at the Q2W schedule, for up to another 12 months. The same treatment guidelines followed during the initial 12-month treatment period will be followed during the retreatment period, including the same dose and frequency of treatments and the same schedule of assessments.
  Interventions: Drug: MEDI4736

INTERVENTIONS:
Drug: MEDI4736 — Patients will be seen the day of administration of MEDI4736. A medical history, with particular reference to toxicities, including medication review, and physical examination will be conducted at each treatment visit.

SUMMARY:
The purpose of this study is to find out what effects, good and/or bad, MEDI4736 has on the patient and cancer.

MEDI4736 is a type of medication called an antibody. Antibodies are normal proteins in the body that help fight infections and possibly cancer. MEDI4736 is a special type of an antibody produced in a laboratory. MEDI4736 works by blocking a specific protein called the Programmed Death Ligand-1 (PDL-1), located on tumor cells.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained.
* Histologically- or cytologically- confirmed CRC.
* Microsatelite-high colorectal cancer (also known as MSI-H, DNA mismatch repair deficient, or sometimes Lynch syndrome); or increased Tumor-Infiltrating Lymphocytes in an archived tumor specimen or fresh biopsy.
* Locally advanced or metastatic CRC
* Subjects have received two or more standard available therapies known to prolong survival and for which they would be considered eligible. At a minimum, such therapies should include regimens containing oxaliplatin and irinotecan in combination with a fluoropyrimidine (e.g., FOLFOX and FOLFIRI or their variants).
* Age ≥ 18 years at time of study entry.
* Eastern Cooperative Oncology Group (ECOG) status of 0 or 1
* Adequate organ and marrow function as defined below:
* Absolute neutrophil count ≥ 1,500/mm3.
* Platelet count ≥ 90,000/mm3.
* AST and ALT ≤ 3 × institutional upper limit of normal (ULN) or ≤ 5 × ULN for subjects with liver metastases.
* Bilirubin ≤ 1.5 × ULN or ≤ 3 × ULN for subjects with documented/suspected Gilbert's disease.
* Serum creatinine ≤ 1.5 x ULN;
* Radiographically measurable disease per RECIST 1.1.
* Life expectancy ≥ 16 weeks.
* Willingness to provide consent for use of archived tissue for research purposes.
* Subjects will be required to agree to a biopsy performed at baseline and again at week 8 of the study in order to be eligible for enrollment in stage 1 of the study
* Females of childbearing potential who are sexually active with a nonsterilized male partner must use 2 methods of effective contraception from screening, and must agree to continue using such precautions for 90 days after the final dose of investigational product; cessation of birth control after this point should be discussed with a responsible physician. Periodic abstinence, the rhythm method, and the withdrawal method are not acceptable methods of birth control.
* Females of childbearing potential are defined as those who are not surgically sterile (ie, bilateral tubal ligation, bilateral oophorectomy, or complete hysterectomy) or postmenopausal (defined as 12 months with no menses without an alternative medical cause).
* Subjects must use 2 acceptable methods of effective contraception as described in below.
* Nonsterilized males who are sexually active with a female partner of childbearing potential must use 2 acceptable methods of effective contraception from Day 1 and for 90 days after receipt of the final dose of investigational product.

Exclusion Criteria:

* Anticancer therapy, monoclonal antibody or major surgery within 4 weeks prior to the first dose of MEDI4736.
* Concurrent use of hormones for non-cancer-related conditions (e.g., insulin for diabetes and hormone replacement therapy) is acceptable.
* Any prior Grade ≥ 3 irAE while receiving immunotherapy (including anti-CTLA-4 or anti-CD137 MAb) or any unresolved irAE of any grade (controlled irAE endocrinopathies are allowed).
* Prior exposure to any anti-PD-1 or anti-PD-L1 antibody.
* Current or prior use of immunosuppressive medication within 28 days before the first dose of MEDI4736, with the exceptions of intranasal and inhaled corticosteroids or systemic corticosteroids at physiological doses, which are not to exceed 10 mg/day of prednisone, or an equivalent corticosteroid.
* Any unresolved toxicity CTCAE >Grade 2 from previous anti-cancer therapy.
* Active autoimmune disease within the past 2 years, except for mild conditions not requiring systemic treatment, such as vitiligo.
* Any concurrent chemotherapy, immunotherapy, biologic or hormonal therapy for cancer treatment. NOTE: Local treatment of isolated lesions, excluding target lesions, for palliative intent is acceptable (e.g., by local ablation, surgery or radiotherapy).
* Active or prior documented inflammatory bowel disease (e.g., Crohn's disease, irritable bowel syndrome, ulcerative colitis).
* Receipt of radiation therapy within 4 weeks prior to starting investigational product, or limited field of radiation for palliation within 2 weeks of the first dose of investigational product.
* Known allergy or reaction to any component of the MEDI4736 formulation or its excipients.
* Known central nervous system (CNS) metastases requiring treatment, such as surgery, radiation or steroids.
* Known history of confirmed primary immunodeficiency.
* History of organ transplant requiring therapeutic immunosuppression.
* Other malignancy within 3 years, except for noninvasive malignancies such as cervical carcinoma in situ (CIS), non-melanomatous carcinoma of the skin or ductal carcinoma in situ (DCIS) of the breast that has/have been surgically cured, or prior malignancy considered by the investigator to be of low likelihood for recurrence.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, active peptic ulcer disease or gastritis, active bleeding diatheses including any patient known to have active hepatitis B, hepatitis C or human immunodeficiency virus (HIV), or psychiatric illness/social situations that would limit compliance with study requirements or compromise the ability of the patient to give written informed consent.
* Women who are pregnant, breast-feeding or male or female patients of reproductive potential who are not employing an effective method of birth control.
* Any other condition(s) that, in the opinion of the investigator, would interfere with evaluation of the investigational product or interpretation of subject safety or study results.
* Subjects who are known to be HIV positive.
* Receipt of live attenuated vaccination within 30 days prior to receiving MEDI4736

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2014-12-02 (Actual); Primary Completion 2020-06-29 (Actual); Study Completion 2020-06-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neil Segal, MD, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Patients With Advanced Colorectal Cancer
Started | 16
Completed | 16
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Patients With Advanced Colorectal Cancer
Number analyzed (Participants) | 16
Age, Continuous [Median (Full Range); unit: years] | 57 [24 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 15
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 12
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 16

OUTCOME MEASURES:

1. Primary Outcome: Best Response Rate
Description: according to RECIST 1.1.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With Advanced Colorectal Cancer
Number analyzed (Participants) | 16
Participants
  Complete Response | 1
  Partial Response | 3
  Stable Response | 4
  Progression of Disease | 4
  Not Entered | 4

2. Secondary Outcome: Number of Participants Evaluated for Toxicities to Determine Safety
Description: Subjects will be evaluated for occurrence of AEs at each visit. Events will be characterized and reported. Safety will also be monitored by performing physical exams and routine laboratory procedures. Terminology Criteria for Adverse Events" V4.0 (CTCAE).
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With Advanced Colorectal Cancer
Number analyzed (Participants) | 16
Participants | 16

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Patients With Advanced Colorectal Cancer
All-Cause Mortality (participants affected / at risk) | 7/16
Serious Adverse Events (participants affected / at risk) | 8/16
Other Adverse Events (participants affected / at risk) | 16/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Patients With Advanced Colorectal Cancer (N=16)
Abdominal pain (Gastrointestinal disorders) | 1
Anorexia (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2
Blood bilirubin increased (Investigations) | 2
Death NOS (General disorders) | 2
Diarrhea (Gastrointestinal disorders) | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
Enterocolitis infectious (Infections and infestations) | 1
Fatigue (General disorders) | 3
Flank pain (Musculoskeletal and connective tissue disorders) | 2
Gait disturbance (General disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Neoplasms ben/mal/unk (inc cyst/polyp) Other, spec (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Non-cardiac chest pain (General disorders) | 1
Small intestinal obstruction (Gastrointestinal disorders) | 2
Tremor (Nervous system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Patients With Advanced Colorectal Cancer (N=16)
Fatigue (General disorders) | 7
Dry skin (Skin and subcutaneous tissue disorders) | 5
Pruritus (Skin and subcutaneous tissue disorders) | 5
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4
Aspartate aminotransferase increased (Investigations) | 3
Diarrhea (Gastrointestinal disorders) | 3
Hyperglycemia (Metabolism and nutrition disorders) | 3
Platelet count decreased (Investigations) | 3
Alanine aminotransferase increased (Investigations) | 2
Anemia (Blood and lymphatic system disorders) | 2
Anorexia (Metabolism and nutrition disorders) | 2
Dizziness (Nervous system disorders) | 1
Dry mouth (Gastrointestinal disorders) | 2
Hyponatremia (Metabolism and nutrition disorders) | 2
Nausea (Gastrointestinal disorders) | 2
Tremor (Nervous system disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 1
Alkaline phosphatase increased (Investigations) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Ataxia (Nervous system disorders) | 1
Blood bilirubin increased (Investigations) | 1
Blurred vision (Eye disorders) | 1
Ear pain (Ear and labyrinth disorders) | 1
Edema limbs (General disorders) | 1
Gait disturbance (General disorders) | 1
Hot flashes (Vascular disorders) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 1
Insomnia (Psychiatric disorders) | 1
Mucositis oral (Gastrointestinal disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
Nervous system disorders - Other, specify (Nervous system disorders) | 1
Peripheral motor neuropathy (Nervous system disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 1
Rash pustular (Infections and infestations) | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1
Syncope (Nervous system disorders) | 1
Urinary frequency (Renal and urinary disorders) | 1
Vomiting (Gastrointestinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-09): https://cdn.clinicaltrials.gov/large-docs/67/NCT02227667/Prot_SAP_000.pdf